CLINICAL TRIAL: NCT04775940
Title: The Use of Perforated Barrier Membranes and IPRF Nano- Micro Sticky Bone in Horizontal Alveolar Ridge Augmentation - Controlled Clinical and Histomorphometric Study
Brief Title: Use of Perforated Barrier Membranes and IPRF Nano- Micro Sticky Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID021701
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Bone Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perforated collagen membrane (Experimental)
  Interventions: Procedure: Perforated collagen membrane
- Occlusive collagen membrane (Active Comparator)
  Interventions: Procedure: Occlusive collagen membrane

INTERVENTIONS:
Procedure: Perforated collagen membrane — Horizontal Bone Augmentation using Perforated Collagen Membrane
  Arms: Perforated collagen membrane
Procedure: Occlusive collagen membrane — Occlusive collagen membrane
  Arms: Occlusive collagen membrane

SUMMARY:
Comparing amount of horizontal bone gain 4 months after alveolar ridge augmentation using IPRF Nano- micro Sticky Bone with perforated collagen membrane versus occlusive barrier membrane by :

1. clinical and Radiographic analysis .
2. Histomorphometric analysis .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult patients.
2. Both sex, males and females. 3-Age from 20 - 40 years old. 4-All patients will be free from any systemic diseases as evidenced by Burkett's oral medicine health history questionnaire.

5-Remaining alveolar bone ≥ 8mm vertically and ≤ 4 mm horizontally. 6-Gingival biotype 1-2mm thickness.

Exclusion Criteria:

1. Smokers.
2. Pregnant and breast feeding females.
3. Mentally retarded Patients.
4. Presence of hematologic disease.
5. Previous radiation, chemotherapy, or immunosuppressive treatments.
6. Diabetes mellitus, metabolic bone disease, ongoing treatment with bisphosphonates drugs, or pregnancy.
7. Anticoagulant drugs, Endocarditis risk factors, renal and hepatic failure

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Horizontal alveolar bone width in mm | 6 months
  Measured By Bone caliber and Cone Beam Computed Tomography (CBCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided